CLINICAL TRIAL: NCT04055415
Title: Safety and Efficacy of Transplantation of Adipose Derived Mesenchymal Stem Cells to Treat Pulmonary Arterial Hypertension
Brief Title: Clinical Study of Adipose Derived Mesenchymal Stem Cells for Treatment of Pulmonary Arterial Hypertension
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liaocheng People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mashengjun2
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension（PH）mesenchymal stem cells(MSC)
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The MSCs of 1×10*6/kg will be given in Central venous catheterization for injection at a total 100 ml . Once every week#a total of two times. The Conventional drug therapy（expectorant，bronchodilator） is used.
  Interventions: Biological: adipose derived mesenchymal stem cells; Drug: Conventional drug therapy（expectorant，bronchodilator）
- Control group (Other): The Conventional drug therapy（expectorant，bronchodilator） is used with the control group
  Interventions: Drug: Conventional drug therapy（expectorant，bronchodilator）

INTERVENTIONS:
Biological: adipose derived mesenchymal stem cells — The MSCs of 1×10*6/kg will be given in Central venous catheterization for injection at a total 100 ml (2) the experimental group was treated with conventional drug and adipose mesenchymal stem cell injection, and adipose MSCs were treated with central venous catheterization. The injection cycle was once every week of two times.Injection dose: 1×106 /kg.
  Arms: Intervention group
Drug: Conventional drug therapy（expectorant，bronchodilator） — Conventional drug therapy（expectorant，bronchodilator）

SUMMARY:
Pulmonary arterial hypertension is a disease characterised by pathological changes in the pulmonary arteries leading to a progressive increase in pulmonary vascular resistance and pulmonary artery pressure. Right ventricular failure is the main cause of death in patients with pulmonary arterial hypertension, and the ability of the right ventricle to adapt to the progressive increase in pulmonary vascular resistance associated with changes to the pulmonary vasculature in pulmonary arterial hypertension is the main determinant of a patient's functional capacity and survival.Mesenchymal stem cells (MSCs)are a subset of adult stem cells residing in many tissues, including bone marrow(BM), adipose tissue, umbilical cord blood. Recent experimental findings have shown the ability of MSCs to home to damaged tissues and to produce paracrine factors with anti-inflammatory properties, potentially resulting in reduction of inflammation and functional recovery of the damaged tissues.It was found that MSCs can significantly improve the pulmonary hemodynamics, lung tissue gross and decrease the pulmonary artery pressure, middle artery thickness and right cardiac hypertrophy by intravenous injection.

ELIGIBILITY:
Inclusion Criteria:

（1）40-75years （2）Male or female （3）The patients that COPD with moderate to severe pulmonary hypertension (pulmonary systolic pressure more than 40mmHg)in relatively stable period （4）To preliminary assess the Patients'lifetime have more than 6 months （5）According to the researchers' judgment, they can abide by the research protocol or Volunteer to participate in the clinical study, understand the study procedure and sign the informed consent in person.

-

Exclusion Criteria:

1. Patients with acute myocardial infarction and cardiac surgery in the past 1 month
2. Surgery may be required within 8 weeks
3. patients with prior pneumonectomy or having acute, chronic pulmonary embolism or other serious pulmonary diseases
4. Having a history of malignant tumor
5. Participated in other clinical investigators in the last 6 months
6. To allergic to penicillin, gentamicin, aminoglycoside, human serum albumin and DMEM medium
7. A woman who is planning to pregnancy, gestation, or lactation
8. Other reasons caused Pulmonary hypertension and heart failure caused by other causes;Severe liver and kidney failure;Autoimmune diseases;Patients with infectious diseases
9. According toThe researchers' judgments, there are concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study
10. According to the researcher's judgment, this study is not suitable for other conditions -

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pulmonary Vascular Resistance from Baseline | Baseline, 4, 12 and 24 weeks

SECONDARY OUTCOMES:
Change from Baseline in Participant Quality of Life Using the SF-36 | Baseline, 4, 12 and 24 weeks
  Eight scale scores are derived from responses to the 36 items of the SF-36 questionnaire which are combined to produce the Physical Component Score and the Mental Component Score. The Physical Component Score is based on the Physical Functioning Scale (10 items), the Role-Physical Scale (4 items), the Bodily Pain Scale (2 items), and the General Health Scale (5 items). The Mental Component Score is based upon the Vitality Scale (4 items), the Social Functioning Scale (2 items), the Role-Emotional Scale (3 items) and the Mental Health Scale (5 items). Each component score is transformed into a 0-100 scale, with higher numbers indicating greater quality of life.
Change in Plasma NT-pro-BNP levels | Baseline, 4, 12 and 24 weeks
  Plasma NT-proBNP concentration is a useful biomarker for PAH as it is associated with changes in right heart morphology and function.
Change in the IL-1β, IL-6, PGE-2, TGF-β, TNF-α and IGF-1 (ng/ul) | Baseline, 4, 12 and 24 weeks
  To assess pre-specified laboratory assessment for change over time with treatment
Incidence of Treatment Adverse | Baseline, 4, 12 and 24 weeks
  An AE was any untoward medical occurrence in a participant
Change in Six Minute Walk distance | Baseline, 4, 12 and 24 weeks
  The 6MWD is a 6 minute walk test. This test, a measure of exercise capacity, assesses the distance that a subject can walk in a period of 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Shengjun Ma, M.D, Study Chair — Liaocheng People's Hospital
Locations (1):
- Liaocheng city people's hospital, Liaocheng, Shandong, China